CLINICAL TRIAL: NCT04729153
Title: Impact of Previous Treatment of HCV Patients by DAADs on Covid-19 Disease Frequency and Severity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Adel Zareh, Doctor, Assiut University
Other Study IDs: DAADs and covid-19
Record Dates: First submitted 2021-01-23; First posted 2021-01-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — 1,4-diacrylateanthracene-9,10-dione

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic HCV patients previously treated by DAADs.
  Interventions: Drug: DAAD Compound
- Chronic HCV patients not treated by DAADs yet.

INTERVENTIONS:
Drug: DAAD Compound — Sofosbuvir , Daclatasvir and ribavirin
  Groups: Chronic HCV patients previously treated by DAADs.

SUMMARY:
Evaluate effect of DAADs on covid-19 disease.

DETAILED DESCRIPTION:
If Chronic HCV patients who already received DAADs are protected against covid 19 and considered to be immune or not And if DAADS can be used in ttt of covid 19

ELIGIBILITY:
Inclusion Criteria:

1. HCV patient with or without LC.
2. >18 years old.
3. Received DAADs at 2019.

Exclusion Criteria:

1. Combined HCV and HIV infected patients.
2. Combined HCV and HBV infected patients.
3. < 18 years old.
4. Pregnant or breast-feeding patients.
5. Patients with autoimmune disease.
6. Patients with multiorgan failure, active cancer, renal insufficiency.
7. Patients received immunosuppressive drugs.
8. Immune compromised patients.
9. Previous confirmed diagnosis of SARS-CoV-2 before starting DAAs.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of DAADs on covid -19 | 12 months (from 1/2/2021 to 1/2/2022)
  If chronic HCV patients who received DAADs suspected to be infected by covid-19 by having findings suggest covid 19 infection in MSCT chest or clinically symptoms or confirmed by nasopharyngeal swab . And if infected what about severity , if they need hospital admission or oxygen therapy or mechanical ventilation ,if they still alive or died